CLINICAL TRIAL: NCT01782703
Title: Defining the Skin and Blood Biomarkers of Pediatric Atopic Dermatitis SUB-STUDY: Defining the Predictive Non-Invasive Biomarkers for Pediatric Atopic Dermatitis (Funded by Regeneron Pharmaceuticals, Inc.)
Brief Title: Defining the Skin and Blood Biomarkers of Pediatric Atopic Dermatitis
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Rockefeller University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Dermatology, Professor of Pediatrics, Northwestern University
Other Study IDs: 2013-15143
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Filaggrin; Biomarkers; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We have retained whole blood and tissue samples (skin and cheek swabs)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Healthy subjects with no history of atopy (atopic dermatitis, asthma, or allergic rhinitis) from 0 months to 17 years of age that are age and sex matched to our atopic dermatitis subjects.
- Atopic Dermatitis: Children with atopic dermatitis from 0 months to 17 years of age.
- Control with Atopy history: Healthy subjects from 0 months to 17 years of age with history of asthma, food allergies, or allergic rhinitis, but no atopic dermatitis or with positive family history of atopy

SUMMARY:
Atopic dermatitis (AD), also known as eczema, is the most common inflammatory skin disorder of children, affecting 10-20% of children and 1-2% of adults.

This skin disorder can be associated with unbearable itchiness and an increased susceptibility to skin infections. The cause of AD is currently poorly understood; therefore, there are no targeted treatment options at present. There have been recent studies in adults with AD that explain the cause and give us new routes to investigate treatment options, however no major studies in this arena have been done in children. We hope to evaluate the skin and blood biomarkers that are found in pediatric AD and compare them to adult AD.

Hypothesis: The immune system worsens the skin barrier issues that are common in atopic dermatitis. We believe there are similar immune and skin abnormalities in adult versus pediatric atopic dermatitis. Finally, blood levels of the activated molecules in atopic dermatitis can serve as surrogates for skin immune activation and will correlate with disease severity.

DETAILED DESCRIPTION:
Objectives:

1. To define the cellular and molecular biomarkers of atopic dermatitis in skin biopsies and blood samples from a pre-adolescent pediatric population and correlate it with disease severity.
2. To measure the skin barrier in atopic dermatitis.
3. To determine quality of life in atopic dermatitis through various questionnaires.

Objectives for the non-invasive biomarkers sub-study:

1. Develop a panel of non-invasive biomarkers in tape strips and serum.
2. Correlate mRNA expression from tape-striped skin with individual markers of severity (EASI, SCORAD, pruritus and TEWL).
3. Correlate mRNA markers in blood with severity scores.
4. Correlate serum protein markers with severity scores.
5. Compare biomarkers based on patient age.
6. Correlate the biomarker candidates from tape strips and blood with the "gold standard" set of biomarkers derived from age-matched skin biopsy samples

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex and must be between the ages of 0 months and 17 years at the time of enrollment (Healthy controls, atopic controls, and AD patients)
* The skin sample and blood sample for healthy controls can have no systemic inflammatory disease or personal or familial history of atopy (hives, food allergy, allergic rhinitis or conjunctivitis, asthma)
* The atopic blood sample controls may have an atopic condition (allergic rhinitis or asthma) but no history of atopic dermatitis
* All controls for skin sampling may have no observable abnormality in the sampled skin and, to further assure the normality of the "normal" skin edges, must not have evidence of inflammation or epidermal change in the lesion to be surgically removed
* AD subjects must have mild to severe atopic dermatitis with either new onset disease within the last 6 months or with acute exacerbation of AD
* Subjects 17 years of age and older and parents/guardians of minors must sign the approved IRB assent and consent form(s) respectively prior to initiation of the study protocol

Exclusion Criteria:

* Subjects unable to give assent or parents unable to give consent due to cognitive delay or inability to understand the assent form either in writing or presented verbally (Healthy controls, atopic controls, and AD patients)
* All subjects whose main diagnosis is deemed unsafe by the study investigator for study participation. Examples include known hemophilia or other blood disorders, or skin infection at the site of blood draw or biopsy (Healthy controls, atopic controls, and AD patients)
* Control subjects with obvious xerosis (Healthy controls and atopic controls)

Ages: 0 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited at Ann and Robert H. Lurie Children's Hospital Dermatology outpatient clinics.
  * 200 children with mild to severe AD, 100 aged-matched and sex-matched healthy (no evidence of atopy) controls, 100 aged-matched and sex-matched controls with an atopic condition (allergic rhinitis or asthma) but no history of atopic dermatitis
  * AD subjects between the ages of 0 months to 4 years of age will be asked to give buccal (cheek) swabs
  * 70 children with mild to severe atopic dermatitis, and 70 age- and sex-matched (but not site-matched) healthy controls (no evidence of atopy), will be enrolled to obtain skin biopsies.
  * 30 children with atopic dermatitis and 30 age/sex matched non-atopic controls for imaging evaluation.
  * Transepidermal water loss values will obtained in 300 healthy controls.
  * Cord blood will be collected from 30 healthy subjects at the time of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cellular infiltrates | One year
  We will examine skin and blood samples for various immune cells known to be involved in atopic dermatitis.
Gene expression | One Year
  We will examine skin and blood samples for various genes known to contribute to atopic dermatitis by analyzing RNA and cytokines.

SECONDARY OUTCOMES:
Correlation of biomarkers to quality of life | One year
  We will analyze the blood and tissue biomarkers to determine whether they are comparable to quality of life and itch (pruritus) measures.

OTHER OUTCOMES:
Development of a panel of non-invasive biomarkers from tape strip samples | Two years
  Development of a panel of non-invasive biomarkers from tape strip samples

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University; Emma Guttman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Northbrook Lurie Children's Outpatient Clinic, Northbrook, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Bieber T. Atopic dermatitis. Ann Dermatol. 2010 May;22(2):125-37. doi: 10.5021/ad.2010.22.2.125. Epub 2010 May 17. PMID 20548901
- [Background] Guttman-Yassky E, Nograles KE, Krueger JG. Contrasting pathogenesis of atopic dermatitis and psoriasis--part II: immune cell subsets and therapeutic concepts. J Allergy Clin Immunol. 2011 Jun;127(6):1420-32. doi: 10.1016/j.jaci.2011.01.054. Epub 2011 Mar 21. PMID 21419481
- [Background] Guttman-Yassky E, Nograles KE, Krueger JG. Contrasting pathogenesis of atopic dermatitis and psoriasis--part I: clinical and pathologic concepts. J Allergy Clin Immunol. 2011 May;127(5):1110-8. doi: 10.1016/j.jaci.2011.01.053. Epub 2011 Mar 8. PMID 21388665
- See also: Eczema: MedlinePlus — http://www.nlm.nih.gov/medlineplus/eczema.html